CLINICAL TRIAL: NCT07265258
Title: A Multicenter, Randomized, Open-Label, Active-Controlled Phase IV Clinical Study to Evaluate the Efficacy and Safety of Teprotumumab N01 in the Treatment of Active Thyroid Eye Disease
Brief Title: A Study of Teprotumumab N01 in Subjects With Active Thyroid Eye Disease
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIBI311A303
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Thyroid Eye Disease
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous glucocorticoid (IVGC) group (Active Comparator)
  Interventions: Drug: Methylprednisolone
- Teprotumumab N01 group (Experimental)
  Interventions: Biological: Teprotumumab N01

INTERVENTIONS:
Biological: Teprotumumab N01 — A total of 8 intravenous infusions of Teprotumumab N01 injection will be adminsitered: 10 mg/kg on Day1, followed by 20 mg/kg in Week3-21, once every 3 weeks(Q3W).
  Arms: Teprotumumab N01 group
Drug: Methylprednisolone — A total of 12 intravenous infusions of methylprednisolone will be administered: 500 mg for the first six doses (on Day 1 and weekly throughout Weeks 1-5), and then 250 mg for the following six doses (weekly throughout Weeks 6-11). Based on disease deterioration and treatment response, participants will receive individualized treatment after IVGC therapy.
  Arms: Intravenous glucocorticoid (IVGC) group

SUMMARY:
This is a multicenter, randomized, open-label, active-controlled Phase IV clinical trial in participants with active thyroid eye disease (TED). Approximately 92 eligible participants will be randomized to the teprotumumab N01 group and the intravenous glucocorticoid (IVGC) group in a 1:1 ratio on Day 1. The randomization stratification factor is diplopia at baseline (Gorman diplopia score ≥1 vs. Gorman diplopia score = 0).

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

1. Written informed consent.
2. Male or female subject between the ages of 18 and 80 years at screening.
3. Weight between 45 kg and 100 kg.
4. Moderate-to-severe active TED:

   * CAS ≥ 3 in the study eye at screening and baseline;
   * Usually associated with at least two of the following: lid retraction ≥ 2 mm, moderate or severe soft tissue involvement, exophthalmos ≥ 3 mm above normal, and/or inconstant or constant diplopia;
   * ≤ 12 months since the onset of active TED symptoms according to subjects' chief complaint or medical record at screening;
5. Exophthalmos ≥ 16 mm in the study eye at baseline.
6. Infertile female participants or fertile female participants with negative blood pregnancy test results during the screening period and agree to take contraceptive measures from screening to 120 days after the last dose; male participants should agree to use contraceptive measures from screening to 120 days after the last dose.

Exclusion Criteria:

Key Exclusion Criteria:

Participants to be excluded (Participants meeting any of the following criteria will be regarded as ineligible):

1. The CAS of the study eye at baseline is reduced by ≥ 2 points compared with that at screening, or the proptosis of the study eye at baseline is reduced by ≥ 2 mm compared with that at screening;
2. Participants previously diagnosed with dysthyroid optic neuropathy (DON), or with DON as determined by the investigator at screening;
3. Patients with corneal ulcers that are not relieved after treatment at the investigator's discretion;
4. Scheduled orbital radiotherapy at any time before baseline or during the study, or surgical treatment for TED, including orbital decompression, strabismus surgery, and eyelid surgery;
5. Participants with poorly controlled thyroid function, defined as free triiodothyronine (FT3) or free thyroxine (FT4) deviating from the normal reference range of the local laboratory by more than 50% at screening;
6. Any other pre-existing disease, metabolic disorder, or physical examination or clinical laboratory abnormality that leads to a reasonable suspicion of a disease or condition that contraindicates the use of the investigational drug, affects the interpretation of study results, or places the participant at high risk of treatment complications;
7. History of tinnitus or other hearing impairment in either ear during the screening period; or abnormal pure tone audiometry results (defined as an average bone conduction hearing threshold of ≥ 25 dB at 0.5, 1, 2, and 4 kHz, or a bone conduction hearing threshold of ≥ 40 dB at any frequency);
8. Poorly controlled diabetes mellitus (defined as glycosylated hemoglobin ≥ 8.0% at screening);
9. Cumulative dose of glucocorticoids used to treat TED ≥ 1 g methylprednisolone equivalents at any time before baseline;
10. Oral or intravenous glucocorticoids within 30 days prior to screening;
11. Peribulbar/periorbital injection of glucocorticoids within 90 days prior to screening;
12. Oral or intravenous administration of any other non-steroidal immunosuppressants within 90 days prior to screening;
13. Use of glucocorticoid eye drops/ointments or use of non-steroidal immunosuppressant eye drops within 30 days prior to screening;
14. Received TEPEZZA or Teprotumumab N01 Injection at any time before screening;
15. Received CD20 antibody or interleukin-6 receptor (IL-6R) antibody at any time before screening;
16. Have received any other TED therapeutic drugs under development (including but not limited to biologics targeting IGF-1R, FcRn, and TSHR) at any time before screening;
17. Use of any other monoclonal antibody within 90 days prior to screening;
18. Female participants in pregnancy or lactation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-09-12 (Estimated); Study Completion 2027-09-04 (Estimated)

PRIMARY OUTCOMES:
The proptosis responder rate of the study eye | Week15
  The proptosis response rate of the study eye was defined as the percentage of participants with a ≥ 2 mm reduction in proptosis of the study eye from baseline and without a ≥ 2 mm increase in proptosis of the fellow eye.
  Proptosis assessment: protrusion of the eye from the orbital rim as measured using a Hertel exophthalmometer.

SECONDARY OUTCOMES:
Change from baseline in proptosis of the study eye | Weeks 15, 24 and 48
  Proptosis assessment: protrusion of the eye from the orbital rim as measured using a Hertel exophthalmometer.
The overall response rate of the study eye | Weeks 15, 24 and 48
  The overall response rate of the study eye was defined as the percentage of participants with a decrease in Clinical Activity Score [CAS] of ≥ 2 points from baseline in the study eye and a decrease in proptosis of ≥ 2 mm from baseline in the study eye, without deterioration in the fellow eye [deterioration is defined as an increase in CAS of ≥ 2 points or an increase in proptosis of ≥ 2 mm].
Change from baseline in proptosis of the study eye on MRI imaging | Week15
  Proptosis of the study eye as measured on orbital MRI imaging.
The proptosis response rate of the study eye | Weeks 24 and 48
  The proptosis response rate of the study eye was defined as the percentage of participants with a ≥ 2 mm reduction in proptosis of the study eye from baseline and without a ≥ 2 mm increase in proptosis of the fellow eye.
The composite effective rate of the study eye | Weeks 15, 24 and 48
  The composite effective rate of the study eye was defined as the percentage of participants with improvement in 2 or more of the 4 indicators [a. ≥2 mm reduction of lid aperture; b. ≥1 point decrease in the five-item CAS (redness of eyelids, swelling of eyelids, redness of conjunctiva, chemosis, and swelling of caruncle or plica); c. ≥2 mm reduction in proptosis; d. ≥8° improvement in ocular motility] in the study eye and without corresponding deterioration in the fellow eye.
Change from baseline in CAS of the study eye | Weeks 15, 24 and 48
  According to the 7-item European Group on Graves' Ophthalmopathy (EUGOGO) amendment, CAS was used to evaluate clinical activity. For each of the following items, one point is given: spontaneous orbital pain, gaze evoked orbital pain, eyelid swelling, eyelid erythema, conjunctival redness, chemosis, and inflammation of caruncle or plica. The sum of these points is the total score, with 0 indicating no clinical activity and 7 indicating the most severe clinical activity.
Rate of CAS of 0 or 1 in the study eye | Weeks 15, 24 and 48
  According to the 7-item European Group on Graves' Ophthalmopathy (EUGOGO) amendment, CAS was used to evaluate clinical activity. For each of the following items, one point is given: spontaneous orbital pain, gaze evoked orbital pain, eyelid swelling, eyelid erythema, conjunctival redness, chemosis, and inflammation of caruncle or plica. The sum of these points is the total score, with 0 indicating no clinical activity and 7 indicating the most severe clinical activity.
The diplopia response rate | Weeks 15, 24 and 48
  The diplopia response rate was defined as the percentage of participants with an improvement in Gorman diplopia score of ≥ 1 grade
The diplopia resolution rate | Weeks 15, 24 and 48
  The diplopia resolution rate was defined as the percentage of participants with Gorman diplopia score = 0
Change from baseline in proptosis of the fellow eye | Weeks 15, 24 and 48
  Proptosis assessment: protrusion of the eye from the orbital rim as measured using a Hertel exophthalmometer.
Change from baseline of the Graves' Ophthalmopathy Quality of Life (GO-QoL) questionnaire score | Weeks 15, 24 and 48
  Change from baseline of the total GO-QoL score, GO-QoL visual functioning subscale and appearance subscale scores
The safety and tolerability of Teprotumumab N01 and IVGC | After receiving Teprotumumab N01 or IVGC treatment for 48 weeks
  Number, incidence, severity, and correlation with the investigational drug or treatment of all ocular and systemic adverse events (AE), treatment-emergent adverse events (TEAE), and serious adverse events (SAE).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China